CLINICAL TRIAL: NCT03744377
Title: Validation ( Endometriosis Health Profile) EHP-30 (Turkish Version) for Patients With Endometriosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: V.K.V. American Hospital, Istanbul (Other)
Responsible Party: Principal Investigator, mehmet ceyhan, Obstetrician and gynecologist, V.K.V. American Hospital, Istanbul
Other Study IDs: VKVAmericanEHP30
Record Dates: First submitted 2018-11-14; First posted 2018-11-16 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: The Endometriosis Health Profile EPH-30 — Self-reported questionnaires

SUMMARY:
Endometriosis can affect quality of life, including physical, psychological and social aspects. It is important to include quality of life measures in evaluating disease severity and response to any given treatment. The 30-item Endometriosis Health Profile (EHP-30) from in-depth interviews with patients with endometriosis is currently the most reliable questionnaire for the measurement of health-related quality of life in women with endometriosis. It includes specific questions addressing the problems faced by patients with endometriosis. The aim of the present study is to validate the Turkish version of EPH 30, a self reported questionnaiere already used internationally, in order to determine the quality of life in women with endometriosis, assess their psychological health and the effectiveness of therapies.

ELIGIBILITY:
Inclusion Criteria:

* Previous surgical and histological diagnosis of endometriosis

Exclusion Criteria:

* Severe underlying comorbidities (gynecological, cardiovascular, respiratory, renal, hematological, endocrine, hepatic, gastrointestinal, neurological)
* Psychiatric diseases
* Refusal or inability to sign the informed consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women referred to Obstetrics and Gynecological Department for the treatment of endometriosis.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-11-15 (Estimated); Primary Completion 2019-07-15 (Estimated); Study Completion 2019-12-15 (Estimated)

PRIMARY OUTCOMES:
Validation of Endometriosis health profile-30 (EHP-30) Turkish version | baseline
  internal consistency and construct validity

CONTACTS AND LOCATIONS:
Locations (1):
- American Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided